CLINICAL TRIAL: NCT00712530
Title: A Phase I Study to Evaluate the Tolerability and Safety of LC002, a DermaVir Vaccine, in HIV-1-infected Subjects Currently Under Treatment With Highly Active Antiretroviral Therapy (HAART)
Brief Title: Single DermaVir Immunization in HIV-1 Infected Patients on HAART
Acronym: GIHU004
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genetic Immunity (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIHU004
Record Dates: First submitted 2008-07-04; First posted 2008-07-10 (Estimated); Results first posted 2013-03-26 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-02

CONDITIONS: HIV Infection
Keywords: HIV; Vaccine; Immune Therapy; DermaVir
MeSH Terms: conditions — HIV Infections | interventions — DermaVir; Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Single low-dose DermaVir immunization
  * 0.1 mg pDNA/subject, 0.8 mL total volume of DermaVir
  * Administered topically with DermaPrep under two skin patches (0.4 mL/patch)
  Interventions: Biological: DermaVir; Drug: HAART
- 2 (Experimental): Single medium-dose DermaVir immunization
  * 0.4 mg pDNA/subject, 3.2 mL total volume of DermaVir
  * Administered topically with DermaPrep under four skin patches (0.8 mL/patch)
  Interventions: Biological: DermaVir; Drug: HAART
- 3 (Experimental): Single high-dose DermaVir immunization
  * 0.8 mg pDNA/subject, 6.4 mL total volume of DermaVir
  * Administered topically with DermaPrep under eight skin patches (0.4 mL/patch)
  Interventions: Biological: DermaVir; Drug: HAART

INTERVENTIONS:
Biological: DermaVir — DermaVir is a synthetic pathogen-like nanomedicine. The active pharmaceutical ingredient is a plasmid DNA expressing fifteen HIV proteins that assemble into HIV-like particles. These particles are safe, cannot replicate, integrate or reverse transcribed. DermaVir is targeted to Langerhans cells with DermaPrep medical device. These DermaVir-containing Langerhans cells migrate to the lymph nodes, where induce HIV-specific cytotoxic T cells that can recognize and kill HIV-infected cells.
  Other Names: LC002
Drug: HAART — Three or more antiretroviral drugs that can fully suppress HIV RNA
  Other Names: Highly active antiretroviral therapy

SUMMARY:
* DermaVir is a plasmid DNA-containing synthetic nanomedicine. It is administered topically with DermaPrep to target Langerhans cells. Langerhans cells with DermaVir migrate to lymph nodes and express HIV-like particles that induce immune responses to kill HIV-infected cells.
* Hypothesis: Single DermaVir immunization is safe and immunogenic measured by induction of HIV-specific precursor/memory T cell responses.
* GIHU004 was a phase I dose escalation study conducted in Hungary. It evaluated the safety and immunogenicity of three dosing regimens of topical DermaVir immunization for the treatment of HIV-infected individuals on fully suppressive highly active antiretroviral therapy (HAART).

DETAILED DESCRIPTION:
This study enrolled nine HIV-infected adult subjects in three sequential dose cohorts. All had durable suppression of HIV-RNA on HAART over the previous 6 months and CD4 count over 300 cells/mm3. Subjects, received on study Day 0 a single DermaVir immunization:

* Low dose: 0.1 mg pDNA, 0.8 mL DermaVir administered under two DermaPrep patches.
* Medium dose: 0.4 mg pDNA, 3.2 mL DermaVir administered under four DermaPrep patches.
* High dose: 0.8 mg pDNA, 6.4 mL DermaVir administered under eight DermaPrep patches.

Subjects were on study for a total of 28 days followed by a post-treatment safety follow-up for 48 weeks. HAART was not interrupted. All subjects completed the 28-day treatment and 48 weeks safety follow up phase.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness of subject or legal guardian/representative to give written informed consent
* HIV-1 infection, as documented by any licensed ELISA test kit and confirmed by Western blot, HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA
* On a stable antiretroviral regimen without changes or interruptions for at least 12 weeks prior to study entry
* Plasma HIV-1 RNA level of less than 50 copies/mL, obtained at least twice within the 12 weeks prior to study entry
* Peak plasma HIV-1 RNA level before initiation of HAART > 1000 copies/mL
* CD4 cell count > 300 cells/mm3 within the 12 weeks prior to study entry
* Nadir (lowest) CD4+ cell count > 250 cells/mm3 at any time prior to study entry
* The following laboratory values, obtained within 30 days prior to study entry:

  * Absolute neutrophil count (ANC) > 1000/mm3
  * Hemoglobin > 9.0 g/dL
  * Platelet count > 50,000/mm3
  * Serum creatinine < upper limit of the laboratory normal range (ULN)
  * AST (SGOT), ALT (SGPT), and alkaline phosphatase < 2.5 x ULN
  * Total bilirubin < 2.5 x ULN
  * Anti-nuclear antibody (ANA) titer of 1:40 or lower and negative for serum anti-double-stranded DNA antibody (anti-ds-DNA) test result at screening.
* All women of reproductive potential must have a negative urine beta-HCG pregnancy test performed within 14 days prior to study entry.
* Female study volunteers who are not of reproductive potential or whose male partner has undergone successful vasectomy are eligible without requiring the use of contraception. Acceptable documentation of menopause, sterilization, and azoospermia is written or oral documentation communicated by clinician.
* All subjects must not participate in a conception process (e.g. active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization) and, if participating in sexual activity that could lead to pregnancy, the study volunteer/ partner must use two reliable methods of contraception simultaneously while receiving the protocol-specified vaccination and for 3 months after the last vaccination.
* Karnofsky performance score > 90 within 30 days prior to study entry
* Men and women age 18-50 years

Exclusion Criteria:

* Viral load measurement > 50 copies/mL within the last 12 weeks prior to study entry
* History of or evidence of active skin disease (e.g. atopic dermatitis), chronic autoimmune disease or any other significant active skin disease
* Treatment with topical corticosteroids in close proximity to the proposed vaccination sites within 2 weeks prior to study entry
* Excessive exposure to the sun (e.g. sunbathing) within 2 weeks prior to study entry
* Use of any local skin treatments to the targeted vaccination sites within 7 days prior to study entry
* History of diabetes and bleeding disorders
* Previous CDC category C event
* Pregnancy or breast-feeding
* Use of immunomodulating therapy, including cyclosporin, IgG-containing products, interleukins, interferons, systemic glucocorticosteroids, or exposure to an experimental HIV vaccine within 6 months prior to study entry
* Receipt of any vaccine within 30 days prior to study entry
* Allergy/sensitivity to study vaccine products, including adhesives, will be excluded
* Active drug or alcohol use or dependence
* Serious illness until subject either completes therapy or is clinically stable on therapy, in the opinion of the site investigator, for at least 14 days prior to study entry
* Hepatitis B surface antigen and/or anti-hepatitis C positive

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2005-01; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denes Banhegyi, MD, Principal Investigator — Saint Laszlo Hospital
Locations (1):
- Saint Laszlo Hospital, Budapest, Budapest, Hungary

REFERENCES:
- [Background] Lorincz O, Toke ER, Somogyi E, Horkay F, Chandran PL, Douglas JF, Szebeni J, Lisziewicz J. Structure and biological activity of pathogen-like synthetic nanomedicines. Nanomedicine. 2012 May;8(4):497-506. doi: 10.1016/j.nano.2011.07.013. Epub 2011 Aug 10. PMID 21839051
- [Background] Somogyi E, Xu J, Gudics A, Toth J, Kovacs AL, Lori F, Lisziewicz J. A plasmid DNA immunogen expressing fifteen protein antigens and complex virus-like particles (VLP+) mimicking naturally occurring HIV. Vaccine. 2011 Jan 17;29(4):744-53. doi: 10.1016/j.vaccine.2010.11.019. Epub 2010 Nov 23. PMID 21109034
- [Background] Toke ER, Lorincz O, Somogyi E, Lisziewicz J. Rational development of a stable liquid formulation for nanomedicine products. Int J Pharm. 2010 Jun 15;392(1-2):261-7. doi: 10.1016/j.ijpharm.2010.03.048. Epub 2010 Mar 25. PMID 20347027
- [Background] Calarota SA, Foli A, Maserati R, Baldanti F, Paolucci S, Young MA, Tsoukas CM, Lisziewicz J, Lori F. HIV-1-specific T cell precursors with high proliferative capacity correlate with low viremia and high CD4 counts in untreated individuals. J Immunol. 2008 May 1;180(9):5907-15. doi: 10.4049/jimmunol.180.9.5907. PMID 18424710
- [Result] Lisziewicz J, Bakare N, Calarota SA, Banhegyi D, Szlavik J, Ujhelyi E, Toke ER, Molnar L, Lisziewicz Z, Autran B, Lori F. Single DermaVir immunization: dose-dependent expansion of precursor/memory T cells against all HIV antigens in HIV-1 infected individuals. PLoS One. 2012;7(5):e35416. doi: 10.1371/journal.pone.0035416. Epub 2012 May 9. PMID 22590502
- [Result] Lisziewicz J, Toke ER. Nanomedicine applications towards the cure of HIV. Nanomedicine. 2013 Jan;9(1):28-38. doi: 10.1016/j.nano.2012.05.012. Epub 2012 May 30. PMID 22659241
- See also: Genetic Immunity's homepage — http://www.geneticimmunity.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nine subjects were sequentially enrolled into each cohort. Participants were recruited from the Szent László Hospital, Budapest, Hungary.
Pre-assignment Details: The first three subjects received a single low-dose DermaVir immunization. Further enrolment of subjects into the medium and high dose cohorts began only after the safety data for cohorts low and medium doses, respectively were available, and the criteria for enrolling into the next cohort were met.
Groups:
- Single Low-dose (0.1 mg pDNA/Subject) DermaVir Immunization: Single low-dose DermaVir immunization
  * 0.1 mg pDNA/subject, 0.8 mL total volume of DermaVir
  * Administered topically with DermaPrep under two skin patches (0.4 mL/patch)
- Single Medium-dose (0.4 mg pDNA/Subject) DermaVir Immunization: Single medium-dose DermaVir immunization
  * 0.4 mg pDNA/subject, 3.2 mL total volume of DermaVir
  * Administered topically with DermaPrep under four skin patches (0.8 mL/patch)
- Single High-dose (0.8 mg pDNA/Subject) DermaVir Immunization: Single high-dose DermaVir immunization
  * 0.8 mg pDNA/subject, 6.4 mL total volume of DermaVir
  * Administered topically with DermaPrep under eight skin patches (0.4 mL/patch)
Period: Overall Study
Arm/Group | Single Low-dose (0.1 mg pDNA/Subject) DermaVir Immunization | Single Medium-dose (0.4 mg pDNA/Subject) DermaVir Immunization | Single High-dose (0.8 mg pDNA/Subject) DermaVir Immunization
Started | 3 | 3 | 3 (Screened 4 patients, but one failed to meet entry criteria due to a history of bleeding and diabetes)
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Low-dose (0.1 mg pDNA/Subject) DermaVir Immunization | Single Medium-dose (0.4 mg pDNA/Subject) DermaVir Immunization | Single High-dose (0.8 mg pDNA/Subject) DermaVir Immunization | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 9
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45 (4.3) | 34 (4.0) | 36 (9.0) | 38 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2
  Male | 2 | 2 | 3 | 7
Region of Enrollment [Number; unit: participants]
  Hungary | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Grade 3 Adverse Event Related to DermaVir Treatment
Description: Occurrence of at least one grade 3 or higher adverse event including signs/symptoms, laboratory toxicities and clinical events possibly, probably or definitely related to study treatment as judged by the Principal Investigator or the site investigators during the 28 days after DermaVir administration.
Time Frame: 28 days
Measure: Number; unit: participants
Arm/Group | Single Low-dose (0.1 mg pDNA/Subject) DermaVir Immunization | Single Medium-dose (0.4 mg pDNA/Subject) DermaVir Immunization | Single High-dose (0.8 mg pDNA/Subject) DermaVir Immunization
Number analyzed (Participants) | 3 | 3 | 3
participants | 0 | 0 | 0

2. Secondary Outcome: CD4+ T Cell Counts/mm3
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: CD4+ T cell counts/mm3
Arm/Group | Single Low-dose (0.1 mg pDNA/Subject) DermaVir Immunization | Single Medium-dose (0.4 mg pDNA/Subject) DermaVir Immunization | Single High-dose (0.8 mg pDNA/Subject) DermaVir Immunization
Number analyzed (Participants) | 3 | 3 | 3
CD4+ T cell counts/mm3 | 893 (461) | 845 (68) | 621 (185)

3. Secondary Outcome: Number of Subjects With Detectable Anti-ds Antibody and ANA
Time Frame: 28 days
Measure: Number; unit: participants
Arm/Group | Single Low-dose (0.1 mg pDNA/Subject) DermaVir Immunization | Single Medium-dose (0.4 mg pDNA/Subject) DermaVir Immunization | Single High-dose (0.8 mg pDNA/Subject) DermaVir Immunization
Number analyzed (Participants) | 3 | 3 | 3
participants | 0 | 0 | 0

4. Secondary Outcome: Number of Subjects Having More Than 50 Copies/mL HIV RNA
Time Frame: 28 days
Measure: Number; unit: participants
Arm/Group | Single Low-dose (0.1 mg pDNA/Subject) DermaVir Immunization | Single Medium-dose (0.4 mg pDNA/Subject) DermaVir Immunization | Single High-dose (0.8 mg pDNA/Subject) DermaVir Immunization
Number analyzed (Participants) | 3 | 3 | 3
participants | 0 | 0 | 0

5. Secondary Outcome: Change in HIV-specific Memory T Cell Responses at Day 28 Compare to Baseline
Description: HIV-specific T cell precursors with high proliferative capacity (PHPC) were quantified as described earlier [Calarota et al. J Immunol 2008]. Gag-, Tat- and Rev-specific T cells were measured representing ca. 25% of HIV epitopes included in DermaVir.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: PHPC count
Arm/Group | Single Low-dose (0.1 mg pDNA/Subject) DermaVir Immunization | Single Medium-dose (0.4 mg pDNA/Subject) DermaVir Immunization | Single High-dose (0.8 mg pDNA/Subject) DermaVir Immunization
Number analyzed (Participants) | 3 | 3 | 3
PHPC count | 325 (266) | 136202 (162287) | 50759 (44792)

6. Other Pre Specified Outcome: Change in HIV-specific Memory T Cell Responses at Week 48
Description: HIV-specific T cell precursors with high proliferative capacity (PHPC) were quantified as described earlier [Calarota et al. J Immunol 2008]. Gag-, Tat- and Rev-specific T cells were measured representing ca. 25% of HIV epitopes included in DermaVir.
  Note, group Single low-dose was measured at 24 weeks, for this group the 48 weeks data is not available
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: PHPC count
Arm/Group | Single Low-dose (0.1 mg pDNA/Subject) DermaVir Immunization | Single Medium-dose (0.4 mg pDNA/Subject) DermaVir Immunization | Single High-dose (0.8 mg pDNA/Subject) DermaVir Immunization
Number analyzed (Participants) | 3 | 3 | 3
PHPC count | 3899 (869) | 9878 (10257) | 18382 (21477)

ADVERSE EVENTS:
Time Frame: From start of study vaccination to study closure
Arm/Group | Single Low-dose (0.1 mg pDNA/Subject) DermaVir Immunization | Single Medium-dose (0.4 mg pDNA/Subject) DermaVir Immunization | Single High-dose (0.8 mg pDNA/Subject) DermaVir Immunization
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 1/3 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Low-dose (0.1 mg pDNA/Subject) DermaVir Immunization (N=3) | Single Medium-dose (0.4 mg pDNA/Subject) DermaVir Immunization (N=3) | Single High-dose (0.8 mg pDNA/Subject) DermaVir Immunization (N=3)
LUMBALGY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Mild, Not related to study medication
FEVER (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) — Mild, related to study medication
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Mild
MYALGIAS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Mild,related to study medication
CHILLS (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) — Mild, related to study medictaion
FATIGUE (General disorders) | 0 (0) | 1 (2) | 0 (0) — Mild
HYPERESTHESY ON THE SITES (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) — Mild
HYPERBILIRUBINAEMY (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) — Moderate
ELEVATED SE BILIRUBIN (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) — Moderate
MACULAR ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Mild, non related to study medication
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Mild

LIMITATIONS AND CAVEATS:
This is a Phase I small sample study that was not powered for the secondary efficacy endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days